CLINICAL TRIAL: NCT04624581
Title: Genetic Characteristics and Determinants of Central Sensitization of Nociception in Fibromylagic Syndrome
Brief Title: FIbromyalgia anD GenetIcs Subgroups (FIDGIS)
Acronym: FIDGIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Service de pharmacologie et toxicologie cliniques, Hôpitaux Universitaire Genève, Rue Gabrielle Perret-Gentil 4, 1205 Genève, SUISSE (Unknown); Association des Fibromyalgiques d'Auvergne, 19 Place de la Résistance, 63800 Cournon d'Auvergne, FRANCE (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RBHP 2020 PICKERING; 2020-A01724-35 (Other: ANSM)
Record Dates: First submitted 2020-11-05; First posted 2020-11-12 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2020-12

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia syndrome; Chronic pain; Widespread pain; genetics; central sensitization
MeSH Terms: conditions — Fibromyalgia; Chronic Pain

STUDY DESIGN:
Intervention Model Description: Exploratory case control pathophysiology study of psychophysical (central sensitization assessment) and genetic (candidate gene panel) characteristics.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient with fibromyalgia syndrome (Experimental): 250 patients with fibromyalgia syndrome (according to American College of Rheumatology 2016) will realize explorations to characterize central sensitization: reflex nociceptive flexion threshold by electrophysiological measure and blood sampling for evaluate the distribution of gene polymorphism.
  Interventions: Device: Electrophysiological measurement of reflex nociceptive flexion threshold (RIII reflex) using Nicolet Vicking device
- Healthy subjects (Sham Comparator): 50 healthy matched volunteers (age, sex and menopausal status for women) will realize explorations to characterize central sensitization: reflex nociceptive flexion threshold by electrophysiological measure and blood sampling for evaluate distribution of gene polymorphism
  Interventions: Device: Electrophysiological measurement of reflex nociceptive flexion threshold (RIII reflex) using Nicolet Vicking device

INTERVENTIONS:
Device: Electrophysiological measurement of reflex nociceptive flexion threshold (RIII reflex) using Nicolet Vicking device — This intervention measures the response to electrical stimulation of the sural nerve using a pair of percutaneous electrodes placed at the external malleolar retro passage of the nerve (2 cm apart) and connected to the stimulation device (Nicolet Vicking). Reflex muscle responses will be collected using surface electrodes placed on the femoral biceps muscle of the participant and connected to an Electromyogram recording device.
  The RIII will be determined twice (rest period between each 10-minute). In order to induce the reflex nociceptive flexion response, repeated cutaneous electrical stimulations (30 to 40) will be applied at the level of the sural nerve following a variable interval of 6 to 10 seconds in order to overcome the phenomena of habituation and predictability. Each stimulus test will consist of a single rectangular pulse of 0.5 ms, of variable intensity (0-100mA) until a reflex nociceptive flexion threshold is detected or a maximum current of 100 mA is reached

SUMMARY:
Fibromyalgia syndrome (FS) is characterized by widespread pain and affect 0.5 to 5 % of the general population, with a higher prevalence in women. Recognized as disease by World Health Organization since 1992, FS concern 1.2 to 2 million of French people and his etiology need to be clarified. This affection is characterized by a higher sensitivity to nociceptive stimulus, articular and muscular pain and associated to: fatigue, headache, sleep disorders, depression and irritated bowel syndrome. The presentation of this symptoms varied according to the patient with a heterogeneity of the clinical, physical, social and psychologic conditions and of the therapeutic responses.

Faced to the heterogeneity of FS, various hypotheses about the development mechanisms exist. Central sensitization could be one of the key mechanisms of FS, it is described as a loss of the natural balance between the transmission of a painful stimulus to the central nervous system and pain-inhibiting mechanisms, which results in permanent or chronic pain.

Moreover, work on the familial character of FS suggests that a genetic component may be involved in its development, but the identification of a genetic determinant is difficult given the multifactorial nature and complexity of FS.

The objective of this study is to characterize the predispositions of central sensitization and genetics in patients with FS compared to a control group, matched in age, sex and menopausal status.

DETAILED DESCRIPTION:
This is an exploratory case control pathophysiology study of psychophysical (central sensitization assessment) and genetic (candidate gene panel) characteristics.

The main objectives of this study are :

Primary: Evaluate the central nociception sensitization characteristics and genetic determinants in fibromyalgic syndrome, comparing a group of patients to matched healthy controls.

Secondary :

* 1) Characterize genetic predispositions of central sensitization in patients with FS compared to matched healthy controls, including confirmation of known genetic markers and potential identification of new genetic variants involved,
* 2) Compare in the area of central sensitization the population of patients with FS and matched healthy controls,
* 3) Compare in the domain of temporal summation the population of patients with FS and matched healthy controls,
* 4) Describe in the clinical field the characteristics of the FS patient population,
* 5) Compare in the areas of quality of life, anxiety/depression and comorbidities, characteristics of the FS patient population and matched healthy controls,
* 6) Compare epigenetic biomarkers of the FS patient population with healthy matched controls,
* 7) Study of the role of the gut microbiota in patients with FS (bio banking)
* 8) Compare in the areas of pain, sound and light sensitivity the population of patients with FS and matched healthy controls.

ELIGIBILITY:
Patient Inclusion criteria :

* Patient between 18 and 65 years old (included),
* Patient with fibromyalgia according to the criteria of the 2016 ACR,
* Patient weighing more than 45kg
* Cooperation and understanding sufficient to comply with the requirements of the study,
* Acceptance to give written consent,
* Affiliation to the French Social Security system,

Patient exclusion criteria :

* treated with antibiotics in the three months prior to inclusion,
* who has reported gastroenteritis in the two months prior to inclusion,
* having a medical and / or surgical history judged by the investigator or his representative to be incompatible with the test
* of childbearing age not using an effective contraceptive method, pregnant or breastfeeding woman.
* participating in another clinical trial, or being in the exclusion period, or having received a total amount of benefits exceeding EUR 4500 over the 12 months preceding the start of the trial,
* benefiting from a measure of legal protection (guardianship, guardianship, deprivation of liberty, safeguard of justice),

Subject inclusion criteria:

* Aged of more than 18 years,
* weighing more than 45kg
* non-painful subjects matched by age (+/- 5 years), by sex, and by menopausal status for women,
* Cooperation and understanding sufficient to comply with the requirements of the study,
* Acceptance of written consent,
* Affiliation to the French Social Security system,
* Registration or acceptance of registration in the National Register of Volunteers participating in research.

Subject exclusion criteria :

* treated with antibiotics in the three months prior to inclusion,
* who has reported gastroenteritis in the two months prior to inclusion,
* Medical and / or surgical history judged by the investigator or his representative to be incompatible with the test,
* Intake of any drugs in the 7 days before inclusion,
* Pregnant or nursing woman
* Participating in another clinical trial, or within the exclusion period, or having received a total amount of compensation in excess of EUR 4500 over the 12 months preceding the start of the trial,
* Benefiting from a measure of legal protection (curatorship, guardianship, safeguard of justice ...)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2022-01-17 (Actual); Study Completion 2022-01-17 (Actual)

PRIMARY OUTCOMES:
Evaluation of nociception flexion reflex (RIII) threshold by electromyography | Day 1
  Patient rested comfortably in a supine position in order to obtain muscular relaxation. Cutaneous electrodes will be applied, and the sural nerve will be stimulated in its retromaleolar track. Electromyographic responses will recorded using the Nicolet Vicking device with a pair of surface electrodes placed over the tendon of the ipsilateral biceps femoris.
  The R-III reflex (objective threshold) will be identified as a multiphasic signal appearing at least 90 ms but less than 250 ms after each stimulation and will be considered to be present when the corrected computed surface was >0.5 mV/ms (positive response).

SECONDARY OUTCOMES:
Evaluation of genetic polymorphism using OpenArray technology | day 1
  Genome-wide association studies highlight that genetic factors are possibly responsible for up to 50% of the disease susceptibility, and several potential candidate genes have been found to be associated to fibromyalgia, including catecholaminergic (COMT), serotoninergic (HTR2A, SLC6A4), dopaminergic (GCH1, TAAR1) and glutamatergic (GRIA4) pathways. The participants will be genotyped for selected SNPs (120 SNPs- OpenArray technology) that have been previously investigated in relation to FM susceptibility, symptoms or potential mechanisms (Algynomics and international publications).
  A single blood sample will be obtained on visit 1 day 1 and 4 aliquotes will be frozen at -80°C and kept frozen until the Open Array Technology analysis
Evaluation of central sensitization | Day 1
  assessed by Central Sensitization Inventory questionnaire
Mechanical temporal summation by numerical scale (0 to 10) | Day 1
  The mechanical temporal summation test will be performed using a 180g (Size 6.45) Von Frey filament applied to the non-dominant arm of the patient/subject who are sitting comfortably in a quiet room. The Von Frey filament will be applied against the skin of the participant at right angle, the manipulator performs a pressure movement until the filament flexes slightly. The participant scores on a numerical verbal scale (0 to 10) the intensity of pain perceived by the application of a single stimulus, and then of ten stimuli
Concise Pain Questionnaire (QCD) | Day 1
  This self-assessment scale allows the patient to characterize the pain in relation to its psychosocial intensity and impact. The patient is asked to answer 9 graduated questions by circling a number from 0 (no pain) to 10 (the most horrible pain you can imagine). Among these questions the patient is asked to blacken the painful areas on a diagram and to put an S if the pain is on the surface or a P if it is deep
Detection of fibromyalgia using the FIRST questionnaire | Day 1
  The FIRST questionnaire is a 6-item self-questionnaire that detects fibromyalgia. The patient is asked to answer "yes" or "no". Five "yes" allow to detect fibromyalgia when pain has persisted for more than 3 months
Evaluation of the impact of fibromyalgia using the FIQ questionnaire | Day 1
  The revised FIQ questionnaire is a 10-item self-questionnaire that assesses the impact of fibromyalgia. The first item is subdivided into 10 questions that assess the impact of the disease in everyday life
Evaluation of the Suspended Symmetrical Dorsal Cellulalgia | Day 1
  The experimenter makes a palpate-roll (by slightly lifting the skin) between the thumb and the other 4 fingers of the hand by following an axis on each side of the patient's spine. The palpate roll begins at the lumbar level and rises to the level of the shoulder blades on each side of the spine. The test is performed on one side of the spine and then on the other. The palpate roll should be performed 5 times on each side of the spine alternately. The investigator should rate for each side and at each pass whether the patient is experiencing pain or not. If the patient does not feel pain after 5 passes, the test is considered negative.
Quality of life by SF-36 quality of life questionnaire | Day 1
  the quality of life of the participants will be assessed by the self-administrated General Questionnaire 36-Item Short Form Survey (SF-36). The SF-36 questionnaire consists of 36 items and assesses an individual's physical and mental health using eleven questions related to eight aspects of health: physical function, role physical, bodily pain, general health, vitality, social function, role emotional, mental health.Global score ranges from 0 to 100.
Emotional status by Hospital Anxiety and Depression scale (HAD) | Day 1
  The Hospital Anxiety and Depression scale is a self-administered questionnaire in 14 items completed by the participant. It is used to determine the levels of anxiety and depression. Seven of the items relate to anxiety and seven relate to depression. Global score ranges from 0 to 42.
Evaluation of micro ARN using OpenArray technology | Day 1
  Studies have shown that thousands of human protein coding genes are regulated by micro RNAs, indicating that micro RNAs are "master regulators" of many important biological processes and some of this microRNA can be implicated in fibromyalgia continuum. The participants micro RNA's will be analyzed for 754 human selected micro RNA (OpenArray technology) that have been previously investigated in relation to FM susceptibility, symptoms or potential mechanisms. A single blood sample will be obtained on visit 1 day 1 and 6 aliquotes will be frozen at -80°C and kept frozen until the Open Array Technology analysis.
Analysis of the microbiota (stool samples), | Day 1
  Identification of bacterial biodiversity by a genetic sequencing analysis of bacterial DNA. The stool samples will be collected and then frozen at -80°C and kept frozen until analysis.
Evaluation of sensitivity to pain by PSQ questionnaire | Day 1
  the sensitivity to pain of the participants will be assessed by the Pain Sensitivity Questionnaire (PSQ). The PSQ questionnaire explore natural sensitivity to pain using questions simulating more or less intense pain situation using 17 questions.
Evaluation of sensitivity to sound by audiometer | Day 1
  the uncomfortable loudness level (ULL) of the participants will be assessed using the procedure of the British audiology society using a conventional audiometer (pure sound emission). The ULL is the level at which the participant responds or clearly feels uncomfortable and confirms this fact after removing the helmet.
Evaluation of sensitivity to light by led panel | Day 1
  the light sensitivity level of the participants will be assessed using a led panel (Lykos Daylight, Manfrotto) in a room without any source of natural light. The light intensity will be progressive (by step of 1 seconds flash light every 20 seconds) and the participant will stop the test when the intensity of the light will be uncomfortable. The light sensitivity is the level at which the participant feels uncomfortable

CONTACTS AND LOCATIONS:
Overall Officials: Gisèle Pickering, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France